CLINICAL TRIAL: NCT04780945
Title: Correlation Between Homologous Recombination Deficiency and Response to Olaparib in Patients With Recurrent Epithelial Ovarian Cancer (EOC)
Brief Title: Functional Analysis of BRCAness
Acronym: FAB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, J.R. Kroep, MD PhD PI, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAB18
Record Dates: First submitted 2019-08-27; First posted 2021-03-04 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Neoplasm Epithelial; Homologous Recombination Deficiency; BRCA1 Mutation; BRCA2 Mutation
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Intervention Model Description: prospective, Dutch, multicenter, single arm phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib monotherapy (Experimental): Patients, irrespective of BRCA status, will be treated with olaparib tablet 300 mg bid
  Interventions: Diagnostic Test: Functional RAD51 assay; Drug: Olaparib Oral Product

INTERVENTIONS:
Diagnostic Test: Functional RAD51 assay — ex vivo functional assay (RAD51 assay also known as Repair Capacity (RECAP) assay ) to test homologous recombination deficiencie (HRD) in viable tumor tissue
  Other Names: RECAP assay
Drug: Olaparib Oral Product — 300 mg bid
  Other Names: Olaparib tablet

SUMMARY:
PARP inhibitors are most effective in homologous recombinant (HR) deficient tumors. There are clear indications that besides BRCA1 or BRCA2 mutated EOC, there is an additional group of EOC having deficiencies in HR (i.e. BRCAness) that might benefit from treatment with PARP inhibitors. Assessment of HR in high grade EOC might therefore serve as a better predictive biomarker and allow the identification of a larger group of patients that could benefit most from platinum based chemotherapy and maintenance treatment with a PARP inhibitor. We recently developed a robust ex vivo functional assay (RAD51 assay;) to test HR in viable tumor tissue. In the proposed study, we will evaluate whether the RAD51 assay predicts sensitivity to therapy with olaparib, in patients with recurrent EOC. With the RAD51 assay we aim to identify a larger number of patients who will benefit from treatment with the PARP inhibitor olaparib than patients with a germline or somatic BRCA mutation only. Furthermore, we aim to identify molecular markers (including genomic markers) that are associated with the outcome of the RAD51 assay. Finally, we will explore whether these molecular markers can be measured in liquid biopsies by analysing ctDNA.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) often presents at an advanced stage, and harbours an unfavourable prognosis. Standard of care includes complete or optimal debulking surgery and chemotherapy, however, most patients experience recurrent disease. Recurrences are often treated with additional chemotherapy, and for selected patients, treatment with PARP inhibitors may be an option. Patients with platinum sensitive recurrent epithelial ovarian cancer (EOC) and a germ-line or somatic BRCA1 or BRCA2 mutation, who are in response to platinum based chemotherapy are currently eligible for maintenance treatment with the Poly (ADP-ribose) polymerase (PARP) inhibitor olaparib after chemotherapy. Germline (11-15%) or somatically acquired (6-7%) BRCA1 and BRCA2 mutations lead to deficiency in homologous recombination (HR) and subsequent less effective DNA repair. PARP inhibitors are most effective in HR deficient tumors. There are clear indications that besides BRCA1 or BRCA2 mutated EOC, there is an additional group of EOC (~15-30%) having deficiencies in HR (i.e. BRCAness) that might benefit from treatment with PARP inhibitors (Mukhopadhyay, Cancer Res 2012; Konstantinopolos, Cancer Discovery 2015; Telli, Clin Cancer Res 2016). Assessment of HR in high grade EOC might therefore serve as a better predictive biomarker and allow the identification of a larger group of patients that could benefit most from platinum based chemotherapy and maintenance treatment with a PARP inhibitor. We recently developed a robust ex vivo functional assay (RAD51 assay;) to test HR in viable tumor tissue (Naipal, Clin. Cancer Res., 2014). It is still unknown however, whether the outcome of the RAD51 assay reliably predicts the sensitivity to platinum-based chemotherapy or PARP inhibitors. In the proposed study, we will therefore evaluate whether the RAD51 assay predicts sensitivity to therapy with olaparib, in patients with recurrent EOC. With the RAD51 assay we aim to identify a larger number of patients who will benefit from treatment with the PARP inhibitor olaparib than patients with a germline or somatic BRCA mutation only. Furthermore, we aim to identify molecular markers (including genomic markers) that are associated with the outcome of the RAD51 assay. Finally, we will explore whether these molecular markers can be measured in liquid biopsies by analysing ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent high grade serous or endometrioid EOC (more than 3 months after platinum containing chemotherapy and unwilling or ineligible for platinum based therapy) with a tumor lesion that is amendable for biopsy or who can undergo ascites drainage prior to treatment.
* Diagnosis of high grade serous or endometrioid EOC confirmed by histology .
* Provision of informed consent prior to any study specific procedures
* Female aged equal or above 18 years
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration olaparib
* Eastern Cooperative Oncology Group performance status 0 to 2
* Patients must have a life expectancy equal or above 16 weeks.
* Postmenopausal or evidence of nonchildbearing status for women of childbearing potential, negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
* Patients willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Evaluable disease, measurable and, or nonmeasurable, that can be accurately assessed at baseline using RECIST by CT or MRI and is suitable for repeated assessment.
* For inclusion in the optional exploratory genetic research and the optional biomarker research, patients must fulfil informed consent for genetic research and informed consent for biomarker research

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last month.
* Any previous treatment with PARP inhibitor, including olaparib.
* Other malignancy within the last 5 years, except, adequately treated nonmelanoma skin cancer, curatively treated in situ cancer, stage 1 and grade 1 endometrial carcinoma, or other solid tumours including breast cancer and lymphomas curatively treated with no evidence of disease for equal or above 3 years.
* Patients receiving radiotherapy within 3 weeks prior to study treatment.
* Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors
* Concomitant use of known strong or moderate CYP3A inducers.
* Persistent toxicities , Common Terminology Criteria for Adverse Event equal or above grade 2, caused by previous cancer therapy, excluding alopecia.
* Patients with symptomatic uncontrolled brain metastases. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active, uncontrolled infection.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Breast feeding women.
* Immunocompromised patients, for example, patients who are known to be serologically positive for human immunodeficiency virus.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with known active hepatitis due to risk of transmitting the infection through blood or other body fluids
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation.
* Patients with myelodysplastic syndrome, acute myeloid leukaemia or with features suggestive of MDS, AML.
* Whole blood transfusions in the last 120 days prior to entry to the study .
* Resting ECG with QTc equal or above 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 55 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 3 years
  The primary endpoint is the RR, defined as the best overall response (partial response and/or complete response) according to RECIST1.1 for both the HR proficient and HR deficient group as determined by the RAD51 assay.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 3 years
  time from start of maintenance olaparib to the date of first documented disease progression or death from any cause, whichever occurs first, of olaparib for the BRCA1 or BRCA2 mutant (germline or somatic) HR deficient group, the non BRCA mutant HR deficient group and the HR proficient group
Overall Survival (OS) | 3 years
  time from start olaparib to death (any cause).
RAD51 test | 3 years
  Percentage of informative RAD51 test results in tumor biopsies and/or ascites
Loss of function mutation | 3 years
  Identify loss of function mutations in genes involved in HR as part of the molecular analysis in the HR proficient and HR deficient group as determined by the RAD51 assay.
NCT-CTC toxicity criteria | 3 years
  Safety and adverse events (AE) of Common Terminology Criteria for Adverse Events version 4.03 (CTCAE) grade 3>5.

OTHER OUTCOMES:
molecular marker in liquid biopsies | 3 years
  molecular marker analysis BRCA/HRD (ctDNA in blood), using NGS and digital PCR analyses

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No